CLINICAL TRIAL: NCT03488394
Title: Phase I/II Study Evaluating Safety and Efficacy of Autologous Hematopoietic Stem and Progenitor Cells Genetically Modified With IDUA Lentiviral Vector Encoding for the Human α-L-iduronidase Gene for the Treatment of Patients Affected by Mucopolysaccharidosis Type I, Hurler Variant
Brief Title: Gene Therapy With Modified Autologous Hematopoietic Stem Cells for the Treatment of Patients With Mucopolysaccharidosis Type I, Hurler Variant
Acronym: TigetT10_MPSIH
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orchard Therapeutics (Industry)
Collaborators: Fondazione Telethon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-514870-29-00
Record Dates: First submitted 2018-03-22; First posted 2018-04-05 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Mucopolysaccharidosis IH
Keywords: Mucopolysaccharidosis IH; Gene Therapy; Transplantation, Autologous; Lentiviral vector
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — Clinical Coding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Gene therapy (autologous, CD34+ cell enriched cells fraction containing HSCs, transduced with the IDUA LV encoding for the human IDUA gene and cryopreserved in cryoformulation medium)
  Interventions: Genetic: Frozen autologous CD34+ hematopoietic stem and progenitor cells genetically modified with the lentiviral vector IDUA LV, encoding for the α-L-iduronidase cDNA, in their final formulation medium.

INTERVENTIONS:
Genetic: Frozen autologous CD34+ hematopoietic stem and progenitor cells genetically modified with the lentiviral vector IDUA LV, encoding for the α-L-iduronidase cDNA, in their final formulation medium. — The drug product target dose is more or equal to 8x10^6 CD34+ cells/Kg, with a minimum dose of 4x10^6 CD34+ cells/Kg and a maximum dose of 35x10^6 CD34+ cells/Kg.
  The product will be injected intravenously.

SUMMARY:
This is a phase I/II study evaluating safety and efficacy of autologous hematopoietic stem and progenitor cells genetically modified with IDUA lentiviral vector encoding for the human α-L-iduronidase gene for the treatment of patients affected by Mucopolysaccharidosis Type I, Hurler variant

DETAILED DESCRIPTION:
Pediatric patients with mucopolysaccharidosis type I will be treated with genetically modified autologous hematopoietic stem cells collected from mobilized peripheral blood (or bone marrow if mobilization is not feasible) and transduced with IDUA lentiviral vector encoding for the human α-L-iduronidase gene.

Patients will be followed for 8 years after gene therapy. After completing participation in this study, subjects will be offered enrollment into an approved long term follow-up (LTFU) study which will enable continued follow-up for up to 15 years post-treatment (per regulatory guidelines for follow up of patients treated with ATMPs).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by parent/legal guardian
* Sex: Males and Females
* Age: ≥ 28 days and ≤ 11 years old
* Biochemically and molecularly proven MPS IH
* Lansky index >80%
* Indication to hematopoietic stem cell transplant
* Lack of a non-heterozygous (for mutated IDUA) HLA-matched sibling donor or a ≥7/8 (4 digits high-resolution typing) HLA-matched cord blood donor with a cellularity ≥5 x 10^7 Total Nucleated Cells (TNC)/Kg after 1-month search.(This criterion will not apply to patients whose country of origin does not offer unrelated donor cord blood transplantation).
* Adequate cardiac, renal, hepatic and pulmonary functions

Exclusion Criteria:

* Use of other investigational agents within 4 weeks prior to study enrolment (within 6 weeks if use of long-acting agents)
* Severe, active viral, bacterial or fungal infection at eligibility evaluation
* Patients affected by neoplasia or family history of familial cancer syndromes
* Cytogenetic alterations associated with high risk of developing hematological malignancies
* History of uncontrolled seizures
* Patients with end-organ damage or any other severe disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Positivity for HIV (serology or RNA), and/or HbsAg and/or HBV DNA and/or HCV RNA and/or Treponema Pallidum or Mycoplasma active infection
* Patients with DQ/IQ <70
* Previous allogeneic hematopoietic stem cells transplantation or gene therapy with a different product
* Contraindications to PeIMP (G-CSF, Plerixafor, Busulfan, Fludarabine, Rituximab)

Ages: 28 Days to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 8 years
  Number and percentage of subjects alive at the end of the trial
Achievement of haematological engraftment | within day +45 after gene therapy
  Percentage of subjects with both neutrophil count more than 500/mm3 and platelets more than 20,000/mm3 (in the absence of platelet transfusion for seven consecutive days) on 3 consecutive blood counts in the first 45 days from ATIMP injection.
Safety of the administration of autologous haematopoietic stem cells transduced with IDUA LV - Short term tolerability | 0-24 hours from ATIMP injection
  Percentage of subjects not experiencing short-term adverse events of any grade and systemic reactions
Safety of the administration of autologous haematopoietic stem cells transduced with IDUA LV - Absence of Replication Competent Lentivirus | Assessed at multiple timepoints up to 8 years post-treatment
  Percentage of subjects without Replication Competent Lentivirus
Safety of the administration of autologous haematopoietic stem cells transduced with IDUA LV - Absence of malignancy or abnormal clonal proliferation | Assessed at multiple timepoints up to 8 years post-treatment
  Percentage of subjects without abnormal clonal proliferation
Overall safety and tolerability (AE) | Assessed at multiple timepoints up to 8 years post-treatment
  The number of AEs (expected/unexpected and/or related/not related) and SAEs (expected/unexpected and/or related/not related) and the percentage of subjects experiencing AEs (expected/unexpected and/or related/not related) and SAEs (expected/unexpected and/or related/not related) will be summarized by severity and within body system involved. Narratives will also be presented. The rate of occurrence of these events will also be estimated.
IDUA activity in blood (up to supraphysiologic levels) at 1-year post-treatment | Assessed at multiple timepoints up to 8 years post-treatment
  IDUA activity measured on peripheral blood dried spot

SECONDARY OUTCOMES:
Anti-IDUA antibody immune response | Assessed at multiple timepoints up to 8 years post-treatment
  Presence or absence and titer of anti-IDUA antibody on serum
Achievement of supraphysiologic IDUA activity in blood | Assessed at multiple timepoints up to 8 years post-treatment
  IDUA activity measured on peripheral blood spots up to supraphysiologic levels as compared with healthy donors. A supraphysiologic IDUA level is defined as >24.31 μmol/L/h, which is the 97.5th percentile of the IDUA distribution in healthy children
IDUA activity in plasma | Assessed at multiple timepoints up to 8 years post-treatment
  IDUA activity measured on plasma samples from peripheral blood.
Engraftment of transduced cells ≥ 0.30 VCN/genome | Assessed at multiple timepoints up to 8 years post-treatment
  Percentage of subjects with engraftment of transduced cells ≥ 0.30 VCN/genome on peripheral blood mononuclear cells (PBMC) and/or bone marrow (BM) progenitor cells.
Normalization of urinary GAGs | Assessed at multiple timepoints up to 8 years post-treatment
  Percentage of subjects achieving normalization of urinary GAG levels (heparan sulfate and dermatan sulfate) measured by HPLC
Normalization of spleen and liver | Assessed at multiple timepoints up to 8 years post-treatment
  Percentage of subjects with normal spleen and liver assessed by clinical examination (palpation) and/or ultrasound
Growth velocity | Assessed at multiple timepoints up to 8 years post-treatment
  length/height for age and cm/year percentiles

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aldenhoven M, Jones SA, Bonney D, Borrill RE, Coussons M, Mercer J, Bierings MB, Versluys B, van Hasselt PM, Wijburg FA, van der Ploeg AT, Wynn RF, Boelens JJ. Hematopoietic cell transplantation for mucopolysaccharidosis patients is safe and effective: results after implementation of international guidelines. Biol Blood Marrow Transplant. 2015 Jun;21(6):1106-9. doi: 10.1016/j.bbmt.2015.02.011. Epub 2015 Feb 20. PMID 25708213
- [Background] Biffi A, Montini E, Lorioli L, Cesani M, Fumagalli F, Plati T, Baldoli C, Martino S, Calabria A, Canale S, Benedicenti F, Vallanti G, Biasco L, Leo S, Kabbara N, Zanetti G, Rizzo WB, Mehta NA, Cicalese MP, Casiraghi M, Boelens JJ, Del Carro U, Dow DJ, Schmidt M, Assanelli A, Neduva V, Di Serio C, Stupka E, Gardner J, von Kalle C, Bordignon C, Ciceri F, Rovelli A, Roncarolo MG, Aiuti A, Sessa M, Naldini L. Lentiviral hematopoietic stem cell gene therapy benefits metachromatic leukodystrophy. Science. 2013 Aug 23;341(6148):1233158. doi: 10.1126/science.1233158. Epub 2013 Jul 11. PMID 23845948
- [Background] Capotondo A, Milazzo R, Politi LS, Quattrini A, Palini A, Plati T, Merella S, Nonis A, di Serio C, Montini E, Naldini L, Biffi A. Brain conditioning is instrumental for successful microglia reconstitution following hematopoietic stem cell transplantation. Proc Natl Acad Sci U S A. 2012 Sep 11;109(37):15018-23. doi: 10.1073/pnas.1205858109. Epub 2012 Aug 23. PMID 22923692
- [Background] Cartier N, Hacein-Bey-Abina S, Bartholomae CC, Veres G, Schmidt M, Kutschera I, Vidaud M, Abel U, Dal-Cortivo L, Caccavelli L, Mahlaoui N, Kiermer V, Mittelstaedt D, Bellesme C, Lahlou N, Lefrere F, Blanche S, Audit M, Payen E, Leboulch P, l'Homme B, Bougneres P, Von Kalle C, Fischer A, Cavazzana-Calvo M, Aubourg P. Hematopoietic stem cell gene therapy with a lentiviral vector in X-linked adrenoleukodystrophy. Science. 2009 Nov 6;326(5954):818-23. doi: 10.1126/science.1171242. PMID 19892975
- [Background] Hong KT, Kang HJ, Kim NH, Kim MS, Lee JW, Kim H, Park KD, Shin HY, Ahn HS. Successful mobilization using a combination of plerixafor and G-CSF in pediatric patients who failed previous chemomobilization with G-CSF alone and possible complications of the treatment. J Hematol Oncol. 2012 Mar 30;5:14. doi: 10.1186/1756-8722-5-14. PMID 22458355
- [Background] Martin HR, Poe MD, Provenzale JM, Kurtzberg J, Mendizabal A, Escolar ML. Neurodevelopmental outcomes of umbilical cord blood transplantation in metachromatic leukodystrophy. Biol Blood Marrow Transplant. 2013 Apr;19(4):616-24. doi: 10.1016/j.bbmt.2013.01.010. Epub 2013 Jan 22. PMID 23348427
- [Background] Montini E, Cesana D, Schmidt M, Sanvito F, Ponzoni M, Bartholomae C, Sergi Sergi L, Benedicenti F, Ambrosi A, Di Serio C, Doglioni C, von Kalle C, Naldini L. Hematopoietic stem cell gene transfer in a tumor-prone mouse model uncovers low genotoxicity of lentiviral vector integration. Nat Biotechnol. 2006 Jun;24(6):687-96. doi: 10.1038/nbt1216. Epub 2006 May 28. PMID 16732270
- [Background] Muenzer J, Fisher A. Advances in the treatment of mucopolysaccharidosis type I. N Engl J Med. 2004 May 6;350(19):1932-4. doi: 10.1056/NEJMp048084. No abstract available. PMID 15128891
- [Background] Shapiro EG, Nestrasil I, Rudser K, Delaney K, Kovac V, Ahmed A, Yund B, Orchard PJ, Eisengart J, Niklason GR, Raiman J, Mamak E, Cowan MJ, Bailey-Olson M, Harmatz P, Shankar SP, Cagle S, Ali N, Steiner RD, Wozniak J, Lim KO, Whitley CB. Neurocognition across the spectrum of mucopolysaccharidosis type I: Age, severity, and treatment. Mol Genet Metab. 2015 Sep-Oct;116(1-2):61-8. doi: 10.1016/j.ymgme.2015.06.002. Epub 2015 Jun 17. PMID 26095521
- [Background] Visigalli I, Delai S, Politi LS, Di Domenico C, Cerri F, Mrak E, D'Isa R, Ungaro D, Stok M, Sanvito F, Mariani E, Staszewsky L, Godi C, Russo I, Cecere F, Del Carro U, Rubinacci A, Brambilla R, Quattrini A, Di Natale P, Ponder K, Naldini L, Biffi A. Gene therapy augments the efficacy of hematopoietic cell transplantation and fully corrects mucopolysaccharidosis type I phenotype in the mouse model. Blood. 2010 Dec 9;116(24):5130-9. doi: 10.1182/blood-2010-04-278234. Epub 2010 Sep 16. PMID 20847202
- [Background] Weisstein JS, Delgado E, Steinbach LS, Hart K, Packman S. Musculoskeletal manifestations of Hurler syndrome: long-term follow-up after bone marrow transplantation. J Pediatr Orthop. 2004 Jan-Feb;24(1):97-101. doi: 10.1097/00004694-200401000-00019. PMID 14676543
- [Background] Wraith JE, Rogers JG, Danks DM. The mucopolysaccharidoses. Aust Paediatr J. 1987 Dec;23(6):329-34. doi: 10.1111/j.1440-1754.1987.tb00284.x. PMID 3124802
- [Derived] Gentner B, Tucci F, Galimberti S, Fumagalli F, De Pellegrin M, Silvani P, Camesasca C, Pontesilli S, Darin S, Ciotti F, Sarzana M, Consiglieri G, Filisetti C, Forni G, Passerini L, Tomasoni D, Cesana D, Calabria A, Spinozzi G, Cicalese MP, Calbi V, Migliavacca M, Barzaghi F, Ferrua F, Gallo V, Miglietta S, Zonari E, Cheruku PS, Forni C, Facchini M, Corti A, Gabaldo M, Zancan S, Gasperini S, Rovelli A, Boelens JJ, Jones SA, Wynn R, Baldoli C, Montini E, Gregori S, Ciceri F, Valsecchi MG, la Marca G, Parini R, Naldini L, Aiuti A, Bernardo ME; MPSI Study Group. Hematopoietic Stem- and Progenitor-Cell Gene Therapy for Hurler Syndrome. N Engl J Med. 2021 Nov 18;385(21):1929-1940. doi: 10.1056/NEJMoa2106596. PMID 34788506